CLINICAL TRIAL: NCT06321679
Title: Response Evaluation of Cancer Therapeutics in Metastatic Castration-Resistant Prostate Cancer (mCRPC) to the Bone: A Whole Body MRI Study
Brief Title: Response Evaluation of Cancer Therapeutics in Metastatic Castration-Resistant Prostate Cancer to the Bone
Acronym: RESPECT
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1269
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: castration-resistant prostate cancer; whole body magnetic resonance imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- WB-MRI: Each patient will undergo imaging with CT, BS and WB-MRI at each study timepoint
  Interventions: Procedure: Imaging evaluation

INTERVENTIONS:
Procedure: Imaging evaluation — each patient will undergo imaging with CT, BS and WB-MRI at each study timepoint

SUMMARY:
This study is aimed to compare whole body MRI (WB-MRI) with Bone Scintigraphy (BS) and Computerized Tomography (CT) scans in patients receiving treatment for metastatic castration-resistant prostate cancer to the bone.

This is a monocentric, prospective observational study.

DETAILED DESCRIPTION:
This is an observational study and will not influence the choice of treatment. The treating clinicians will be able to use any clinical treatment regimen that is considered appropriated for the patient. This may include hormonal therapy or chemotherapy or therapy with radium-223. In addition, patients may be treated with bisphosphonates/denosumab, and granulocity-colony stimulating factor. The duration of therapy, doses, schedules, timing, premedication, patient monitoring during treatment, dose adjustments, and duration of therapy are entirely at the discretion of the treating clinician.

The use of radiotherapy is permitted, but the details including fields used must be communicated to the reporting radiologist to ensure this does not affect the interpretation of imaging. All other supportive or palliative treatments are permitted.

All patients will undergo imaging assessments as follows:

* At baseline, CT, BS (99mTc-MDP) and Whole Body-Magnetic Resonance Imaging (WB-MRI) will be performed.
* Follow-up imaging will be CT, BS and WB-MRI performed every 12 weeks until week 96, and then every 24 weeks until disease progression occurs or week 192.

Additional patient assessments to be performed include:

* questionnaires at baseline, week 36 and end of study to evaluate patient perception, acceptance and preferences regarding the imaging modalities.
* clinical and physical examinations according to routine clinical practice. The radiologist reporting the WB-MRI will be blinded to the results of the CT and BS.

The radiologist reporting the CT and the nuclear medicine physician reporting the BS will likewise be blinded to the results of the WB-MRI.

Neither treating clinicians nor patients will be blinded at any point.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of castration-resistant prostate cancer,
* Single or multiple bone metastases,
* Life expectancy of over 6 months,
* No current active malignancy other than prostate cancer,
* Provision of written informed consent.

Exclusion Criteria:

* Absolute contraindication to WB-MRI, CT or BS,
* Radical treatment of sole site of metastatic disease (e.g. Cyberknife to solitary metastatic lesion),
* Psychological, familial, sociological or geographical conditions that would hamper compliance with the study protocol; such conditions are to be discussed with the patient as part of the informed consent process.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The estimated rate of recruitment to the study 6-7 patients a month, thus it is expected that patient accrual will be completed within 7 months.
  Based on recent treatment patterns, the expected distribution of treatments is:
  * Hormonal treatments
    * Enzalutamide: 14 patients
    * Abiraterone: 8 patients
  * Chemotherapy
    * Docetaxel: 11 patients
    * Cabazitaxel: 5 patients
  * Radiopharmaceutical drug - Radium-223: 2 patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression in bone metastasis identify by WB-MRI | 192 weeks
  the proportion of WB-MRI examinations that identify disease progression in bone metastases prior to CT + BS

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Petralia, Principal Investigator — European Institute of Oncology
Locations (1):
- IEO Istituto Europeo di Oncologia, Milan, Italy